CLINICAL TRIAL: NCT01436747
Title: Efficacy and Safety of Selective Vitamin D Receptor Activation With Paricalcitol for Reduction of Proteinuria in Kidney Transplant Recipients: a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Paricalcitol for Reduction of Proteinuria in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Miha Arnol, M.D., Ph.D., Miha Arnol, M.D., Ph.D., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31-06-2011
Record Dates: First submitted 2011-09-14; First posted 2011-09-20 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Disorder of Transplanted Kidney; Proteinuria; Albuminuria
Keywords: Kidney transplantation; Proteinuria; Albuminuria; Vitamin D; Paricalcitol
MeSH Terms: conditions — Proteinuria; Albuminuria | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol (Active Comparator)
  Interventions: Drug: Paricalcitol
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — 2 micrograms daily, peroral, 24 weeks
  Other Names: Zemplar
  Arms: Paricalcitol
Drug: Placebo — 2 micrograms daily, peroral, 24 weeks
  Arms: Matching placebo

SUMMARY:
The study 'Safety and Efficacy of Paricalcitol for Reduction of Proteinuria in Kidney Transplant Recipients' is designed to assess the effects of paricalcitol in kidney transplant recipients with proteinuria.

It is a single centre, randomized, placebo-controlled, double-blind clinical trial that tests the hypothesis that 24 weeks' treatment with paricalcitol compared to placebo will result in a decrease in urinary protein excretion in recipients of a kidney transplant at least three months after transplantation. Additionally, the effects of paricalcitol on albuminuria, estimated glomerular filtration rate, and blood pressure will be investigated.

DETAILED DESCRIPTION:
Kidney transplantation is the treatment of choice for end-stage renal disease patients. In comparison to dialysis it offers longer survival and better quality of life to certain patients with end stage renal disease. In the last two decades, short-term (i.e. 1- and 3-year) kidney transplant survival has increased significantly and is currently exceeding 90% in state-of-the-art transplant centers. This is considered to be due to the safe and effective immunosuppressive therapy in the early post-transplant period, and to the careful management of patients with chronic renal disease (CRD) before and after the transplantation. In spite of the progress described above, long-term (i.e. 5- and 10-year) transplant survival has not significantly improved over the recent decades. Two main causes for long-term loss of transplanted kidneys are the development of the transplant chronic kidney disease (CKD) (i.e. chronic allograft nephropathy) and patient death with a functioning transplant due to cardiovascular events.

Proteinuria (> 150 mg of proteins in urine per day) is a manifestation of kidney disease and is an important risk factor for CKD progression. This applies also to kidney transplant recipients. Studies have shown that proteinuria is present in 20-40% of transplanted patients. According to observational studies, proteinuria is an independent predictor for CKD progression and transplant failure, as well as of increased risk for cardiovascular events. In CKD patients, treatment with renin-angiotensin-aldosterone system inhibitors (RAAS - angiotensin converting enzyme inhibitors, angiotensin receptor blockers, aldosterone receptor blockers) reduces proteinuria and thus slows the renal disease progression. In spite of the demonstrated renoprotective effect of RAAS inhibitors, the risk for CKD progression remains high. Furthermore, large epidemiological studies have not shown clinically significant effect of RAAS inhibitor therapy on the reduction of cardiovascular risk. In spite of an optimal RAAS inhibitor therapy, renal and cardiovascular diseases continue to progress, which is also associated with persistent proteinuria. Therefore, new treatment modalities to reduce proteinuria with consequent delay in the progression of CKD and cardiovascular disease are being sought.

Calcitriol is an active form of vitamin D produced in the kidneys. It is important for calcium and phosphate metabolism, as well as for bone mineralization. Decreasing blood calcitriol levels are associated with declining renal function. Decreased calcitriol levels in patients with CKD contribute to the development of secondary hyperparathyroidism. Furthermore, calcitriol deficiency is associated with increased proteinuria and further progression of renal impairment. Vitamin D deficiency in patients with end stage renal disease is also related to higher cardiovascular mortality. The pleiotropic effects of calcitriol probably reflect the presence of vitamin D receptors in different tissues; it is via these receptors that calcitriol exerts its pharmacological effects. Vitamin D receptors have been found not only in kidneys and bones, but also in the cells of the myocardium, in the vascular endothelium, the endocrine part of the pancreas, the intestine and the prostate.

Treatment with an analogue of the active vitamin D form, paricalcitol, significantly reduced proteinuria and slowed progression of renal disease in animal models as well as in patients with CKD, particularly in patients diabetes and diabetic nephropathy. This is considered to be due to the positive effect of paricalcitol on RAAS inhibition in the kidneys, which is independent of calcium and parathormone metabolism. Reduced proteinuria leads to a reduced inflammatory response, preservation of the glomerular basement membrane structure and slowing of glomerulosclerosis.

The positive effects of paricalcitol on the reduction of proteinuria observed in patients with CKD may also be important for kidney transplant recipients: by reducing the proteinuria, progression of CKD in the transplanted kidney might be delayed and the risk for cardiovascular events reduced. This might contribute to the improvement of long-term kidney transplant survival, which has not changed significantly in the last two decades.

This study tests the hypothesis whether paricalcitol persistently reduces proteinuria in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a deceased donor kidney transplant at least 3 months after transplantation
* Urinary protein to creatinine ratio (UPCR) > 200 mg/g (20 mg/mmol) as determined by the the mean of three second morning void urine specimens
* Subject is on stable immunosuppression for at least 3 months
* Subject is on stable doses of antihypertensive medications for at least 3 months
* Subject is not expected to begin dialysis for at least 6 months
* Estimated glomerular filtration rate > 15 ml/min/1.73 m2
* Corrected serum calcium level < 2.6 mmol/l
* Intact parathormone value > 30 pg/ml

Exclusion Criteria:

* Subjects on vitamin D receptor activation therapy within 3 months prior to the first study visit
* Acute kidney injury within 3 months of the first study visit
* Subjects with poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The percentage change in urinary protein to creatinine ratio (UPCR) from baseline to the last measurement during treatment. | baseline and 6 months

SECONDARY OUTCOMES:
The percentage change in urinary albumin to creatinine ratio (UACR) from baseline to the last measurement during treatment. | baseline and 6 months
Change in 24-hour urinary protein excretion form baseline to the last measurement during treatment. | baseline and 6 months
The proportion of patients achieving at least a 15 mg/mmol reduction in the last on-treatment UPCR level from the baseline. | baseline and 6 months
Change in estimated glomerular filtration rate, blood pressure and biomarkers, including (but not limited to) C-reactive protein, plasma renin activity, aldosterone. | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miha Arnol, M.D., Ph.D., Principal Investigator — University Medical Centre Ljubljana, Department of Nephrology; Aljoša Kandus, M.D., Ph.D., Study Chair — University Medical Centre Ljubljana, Department of Nephrology
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Oblak M, Mlinsek G, Kandus A, Buturovic-Ponikvar J, Arnol M. Paricalcitol versus placebo for reduction of proteinuria in kidney transplant recipients: a double-blind, randomized controlled trial. Transpl Int. 2018 Dec;31(12):1391-1404. doi: 10.1111/tri.13323. Epub 2018 Aug 20. PMID 30062716